CLINICAL TRIAL: NCT04700891
Title: Correlation of Preoperative Olfactory Identification Function With Preoperative Frailty and With Postoperative Complications and Mortality Following Elective Surgery
Brief Title: Correlation of Preoperative Olfactory Identification Function With Frailty and Postoperative Complications and Mortality
Acronym: POOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020/22JAN/050
Record Dates: First submitted 2020-12-18; First posted 2021-01-08 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Frailty; Perioperative/Postoperative Complications; Olfactory Disorder
MeSH Terms: conditions — Frailty; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled for elective surgery aged 65 and + (Experimental)
  Interventions: Diagnostic Test: Olfactory identification test; Diagnostic Test: Edmonton Frail Scale; Diagnostic Test: Handgrip strength

INTERVENTIONS:
Diagnostic Test: Olfactory identification test — Burghart Sniffin' Sticks "Screening 12 Test" Olfactory function will be evaluated through the Sniffin' Sticks test which is a validated psychophysical testing method. Sniffin' Sticks test is based on pen-like odor dispensing devices that will be presented to the patients. The short version of this test will be used and will consist solely of a test of odor identification function.
Diagnostic Test: Edmonton Frail Scale — The Edmonton Frail Scale (EFS) involves nine domains of frailty : functional performance, cognitive function, general health, functional independence, social support, used medications, nutrition, mood and continence. It has been validated with respect to comprehensive geriatric assessment and to other screening tools related to frail state. EFS test is considered most appropriate for use in routine preoperative screening and only requires 5 minutes.
Diagnostic Test: Handgrip strength — Handgrip strength is a simple and reliable measurement technique for the assessment of maximal voluntary hand force. Handgrip strength is used as a reflect of nutritional status and muscle mass, physical function and health status. Measurement will be realized using a digital handgrip dynamometer. Patients will be asked to grip the dynamometer with the second finger node at 90° angle to the handle and to grab the handle as strongly as they can. Maximal grip strength will be checked with the forearm away from the body in standing position.

SUMMARY:
The aim of this research project is to evaluate whether olfactory identification impairment is a reliable predictor of preoperative frailty and of postoperative complications and mortality in a population of older patients scheduled for elective surgery.

1. The investigators will measure preoperative olfactory identification function and evaluate whether olfactory impairment predicts frailty, using the Edmonton Frail Scale and handgrip strength.
2. The investigators will analyze whether preoperative olfactory impairment predicts postoperative complications and mortality.

DETAILED DESCRIPTION:
Olfactory impairment increases with age, affecting more than 50% of the population aged between 65 and 80 years old. Recently, many studies have demonstrated a strong association between olfactory impairment and overall mortality risk. At the moment, the underlying physiopathology linking olfactory impairment to mortality remains unknown and only putative mechanisms are suggested.

Among them, accelerated physiological brain aging seems to be involved, making olfactory decline a possible marker of frailty. To date, only a few studies (mostly using subjective olfactory assessment) investigated the potential relationship between olfactory impairment and frailty. Surgery, and more broadly the perioperative period, remains a major source of morbidity and mortality. Meanwhile, the average age of the surgical population continues to rise, making preoperative risk assessment an essential step in order to detect the most vulnerable patients. Yet, it is well-known that frailty is associated with worse perioperative outcome. The first objective of this research project is thus to evaluate olfactory identification function of preoperative older surgical patients in light of an assessment of their frailty status. Frailty will be tested with the Edmonton Frail Scale and handgrip strength, which are both validated tools. The second objective is to correlate postoperative morbidity and mortality with preoperative olfactory function. Hopefully, this research project will address the misunderstood link between olfactory impairment and mortality, focusing on frailty assessment and using surgery as a heavy stressor for the older patient.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery (covering general, gynecologic, urologic, orthopedic, plastic, head and neck, spine neurosurgery)

Exclusion Criteria:

* Day case surgery
* History of neurological or psychiatric disorder
* History of severe head trauma
* History of olfactory trouble or chronic rhinosinusitis or sinus surgery
* History of suspected or diagnosed COVID-19

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 167 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of frailty | The day before surgery (preoperative period)
  Analysis of the prevalence of frailty (assessed by the Edmonton Frail Scale and handgrip strength) according to preoperative olfactory identification function
Incidence of postoperative complications and mortality | Up to 1 year postoperatively
  Analysis of the incidence of postoperative complications and mortality according to preoperative olfactory identification function

OTHER OUTCOMES:
Postoperative olfactory identification function | During first postoperative day
  Comparison of preoperative and postoperative olfactory identification function (assessed by the Sniffin' Sticks "Screening 12 test")

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Van Regemorter, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pinto JM, Wroblewski KE, Kern DW, Schumm LP, McClintock MK. Olfactory dysfunction predicts 5-year mortality in older adults. PLoS One. 2014 Oct 1;9(10):e107541. doi: 10.1371/journal.pone.0107541. eCollection 2014. PMID 25271633
- [Background] Schubert CR, Fischer ME, Pinto AA, Klein BEK, Klein R, Tweed TS, Cruickshanks KJ. Sensory Impairments and Risk of Mortality in Older Adults. J Gerontol A Biol Sci Med Sci. 2017 May 1;72(5):710-715. doi: 10.1093/gerona/glw036. PMID 26946102
- [Background] Van Regemorter V, Hummel T, Rosenzweig F, Mouraux A, Rombaux P, Huart C. Mechanisms Linking Olfactory Impairment and Risk of Mortality. Front Neurosci. 2020 Feb 21;14:140. doi: 10.3389/fnins.2020.00140. eCollection 2020. PMID 32153360
- [Background] Somekawa S, Mine T, Ono K, Hayashi N, Obuchi S, Yoshida H, Kawai H, Fujiwara Y, Hirano H, Kojima M, Ihara K, Kim H. Relationship between Sensory Perception and Frailty in a Community-Dwelling Elderly Population. J Nutr Health Aging. 2017;21(6):710-714. doi: 10.1007/s12603-016-0836-5. PMID 28537337
- [Background] Laudisio A, Navarini L, Margiotta DPE, Fontana DO, Chiarella I, Spitaleri D, Bandinelli S, Gemma A, Ferrucci L, Incalzi RA. The Association of Olfactory Dysfunction, Frailty, and Mortality Is Mediated by Inflammation: Results from the InCHIANTI Study. J Immunol Res. 2019 Feb 20;2019:3128231. doi: 10.1155/2019/3128231. eCollection 2019. PMID 30915369
- [Background] Harita M, Miwa T, Shiga H, Yamada K, Sugiyama E, Okabe Y, Miyake Y, Okuno T, Iritani O, Morimoto S. Association of olfactory impairment with indexes of sarcopenia and frailty in community-dwelling older adults. Geriatr Gerontol Int. 2019 May;19(5):384-391. doi: 10.1111/ggi.13621. Epub 2019 Apr 9. PMID 30968523
- [Derived] Van Regemorter V, Coulie R, Dollase J, Momeni M, Stouffs A, Quenon L, Mouraux A, Huart C. Poor preoperative performance at Clock Drawing Test is associated with postoperative decline in olfaction in older patients: an observational pilot study. BMC Anesthesiol. 2023 Aug 30;23(1):295. doi: 10.1186/s12871-023-02256-0. PMID 37648990